CLINICAL TRIAL: NCT04361942
Title: Double Blind, Placebo-controlled, Phase I/II Clinical Trial to Evaluate Safety and Efficacy of Allogeneic Mesenchymal Stem/Stromal Cells MSV-allo for Treatment of Acute Respiratory Failure in Patients With COVID-19 Pneumonia (MSV-COVID)
Brief Title: Treatment of Severe COVID-19 Pneumonia With Allogeneic Mesenchymal Stem Cells
Acronym: MSV-COVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Red de Terapia Celular (Industry)
Collaborators: Citospin (Industry); University of Valladolid (Other); Castilla-León Health Service (Other); Hospital del Rio Hortega (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TerCel_007; 2020-001682-36 (EudraCT Number)
Record Dates: First submitted 2020-04-17; First posted 2020-04-24 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19; Mesenchymal Stromal Cells; Mesenchymal Stem Cells; MSV
MeSH Terms: conditions — COVID-19 | interventions — Genes, mos; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both experimental and placebo groups will receive a similar endovenous injection with either cells or placebo, respectively. Blind to participant, investigator and care providers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal Stem Cells (MSCs) (Experimental): Intravenous injection of 1 million MSCs (MSV cells)/Kg suspended in 100 ml of physiological saline solution.
  Interventions: Biological: Mesenchymal Stem Cells (MSCs)
- Placebo (Placebo Comparator): Intravenous injection of 100 ml of physiological saline solution containing no cells
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Mesenchymal Stem Cells (MSCs) — Intravenous injection of 1 million MSCs (MSV cells)/Kg suspended in 100 ml physiological saline solution.
  Other Names: MSV (GMP-compliant MSCs manufactured by IBGM in Valladolid)
  Arms: Mesenchymal Stem Cells (MSCs)
Other: Placebo — Intravenous injection of 100 ml physiological saline solution containing no cells
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Novel coronavirus disease COVID-19, produced by SARS-CoV-2, has become a health emergency around the world. Since first patients were detected in Wuhan (China), in December 2019, COVID-19 has spread quickly worldwide, being a severe threat to public health. Fever, dry cough, shortness of breath and breathing distress are the main characteristics of COVID-19 infection. Some patients develop overwhelming lung inflammation and acute respiratory failure, for which there is no specific therapy. Therefore, safe and effective treatment for COVID-19 pneumonia is utterly necessary, mainly in critical cases. Mesenchymal stem/stromal cells (MSCs) have been widely used in the immune-mediated inflammatory diseases. MSCs can regulate both innate and adaptive immunity by suppressing the proliferation, differentiation and activation of different cells. These immunomodulatory properties of MSCs support performance of the double-blind, placebo-controlled, randomized, phase I/II clinical trial to evaluate safety and efficacy of allogeneic MSCs for treatment of severe COVID-19 pneumonia.

DETAILED DESCRIPTION:
Novel coronavirus disease COVID-19, produced by SARS-CoV-2, has spread quickly from Wuhan (China) to worldwide. On April 15, 2020, the World Health Organization (WHO) has reported 1.914.916 confirmed cases and 123.010 deaths globally, being a severe threat to public health.

Some patients develop overwhelming lung inflammation and acute respiratory failure. Several reports demonstrated that SARS-CoV-2 specifically recognize the angiotensin I converting ezyme 2 receptor (ACE2) and ACE2-positive cells are infected by the virus. ACE2 receptor is widely present on the human cells surface such as alveolar type II cells and capillary endothelium, among others. SARS-CoV-2 infects cells and stimulates a terrible cytokine storm in the lung followed by edema, dysfunction of the air exchange and acute respiratory distress which may lead to death. Further, once SARS-CoV-2 enters in blood circulation, it can easily spread to some systems and organs, causing significant damage. Under these circumstances, it is reasonable to believe that the inhibition of inflammatory response is the key to treat COVID-19 pneumonia.

Mesenchymal stem/stromal cells (MSCs) have been widely used in the immune-mediated inflammatory diseases. MSCs can regulate both innate and adaptive immunity by suppressing the proliferation, differentiation and activation of different cells. Some studies have shown that MSCs can significantly reduce acute lung injury in mice caused by H9N2 and H5N1 viruses, reducing proinflammatory cytokines and inflammatory cells into the lungs.

These immunomodulatory properties of MSCs support performance of the placebo-controlled, double-blind (neither the participant nor the investigator will know if active drug or placebo is assigned), randomized (assigned by chance), phase I/II clinical trial in which subjects with severe COVID-19 pneumonia will receive either MSCs (1 million cells/kg) or placebo by intravenous injection. The administration of cells will be done only once.

ELIGIBILITY:
Inclusion Criteria:

1. Women or men of ≥ 18 years of age
2. SARS-CoV-2 infection confirmed by molecular testing.
3. Admitted to the Intensive Care Unit with pneumonia by COVID-19 infection and intubated in the last 48 hours, that meet at least one of these criteria:

   1. Respiratory distress.
   2. Respiratory rate (RR) ≥ 30 rpm.
   3. Basal oxygen saturation at rest ≤ 93%.
   4. Arterial partial pressure of oxygen (PaO2) / inspiratory fraction of oxygen (FiO2) ≤ 300 mmHg.
4. Consent of the patient or his/her legal representative for participation in the study.

Exclusion Criteria:

1. Active tumor disease.
2. Pregnancy.
3. Participation in another active clinical trial.
4. Any circumstance that in the researcher's opinion justifies the patient's non-participation in the trial.
5. Not consent to participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in whom removal of invasive mechanical ventilation (IMV) has been achieved | 0-7 days
  Index of therapy success to preserve Intensive Care Unit (ICU) space.
Overall survival | 0-28 days
  To measure global success

SECONDARY OUTCOMES:
Complete clinical response | 0-Event/Loss to follow-up
  Proportion of patients over time that meet the weaning criteria, defined as (i) PaO2/FiO2 ≥ 200 mmHg, (ii) mechanical ventilation with PEEP ≤ 8 (only if BMI<30), (iii) mechanical ventilation with FiO2 ≤ 50% and (iv) no continuous relaxation (cisatracurium) or prone maneuvers in the last 24 hours.
Complete radiological response | 0-28 days
  Proportion of patients over time that show lung images free from opacities or condensations
Radiological improvement of pulmonary images | 0-5 days
  Change in the proportion of lung sections affected by opacities/condensations in chest X-ray images
Removal of invasive mechanical ventilation (IMV) | 0-28 days
  Proportion of patients over time that reach the event (removal of IMV)

OTHER OUTCOMES:
Levels of cytokines and other inflammatory markers in peripheral blood | 0-7 days
  Interleukin-6 (IL-6), D dimer, C reactive protein (CRP), lactate dehydrogenase (LDH), procalcitonin.
Levels of circulating immune cells | 0-7 days
  B cells, NK cells, T cells, CD4+ T cells, CD8+ T cells
Levels of renal and liver function markers | 0-7 days
  Urea, creatinine, gamma-glutamyltransferase (GGT), glutamate-pyruvate transaminase (GPT), glutamate-oxalacetate transaminase (GOT).

CONTACTS AND LOCATIONS:
Overall Officials: Julia Barbado, MD, PhD, Study Chair — University Hospital Río Hortega, Valladolid, Spain; Rosa Conde, PhD, Study Director — University Hospital Río Hortega, Valladolid, Spain; Margarita González-Vallinas, PhD, Principal Investigator — University of Valladolid
Locations (1):
- Hospital Universitario Rio Hortega, Valladolid, Spain

REFERENCES:
- [Background] Vega A, Martin-Ferrero MA, Del Canto F, Alberca M, Garcia V, Munar A, Orozco L, Soler R, Fuertes JJ, Huguet M, Sanchez A, Garcia-Sancho J. Treatment of Knee Osteoarthritis With Allogeneic Bone Marrow Mesenchymal Stem Cells: A Randomized Controlled Trial. Transplantation. 2015 Aug;99(8):1681-90. doi: 10.1097/TP.0000000000000678. PMID 25822648
- [Background] Noriega DC, Ardura F, Hernandez-Ramajo R, Martin-Ferrero MA, Sanchez-Lite I, Toribio B, Alberca M, Garcia V, Moraleda JM, Sanchez A, Garcia-Sancho J. Intervertebral Disc Repair by Allogeneic Mesenchymal Bone Marrow Cells: A Randomized Controlled Trial. Transplantation. 2017 Aug;101(8):1945-1951. doi: 10.1097/TP.0000000000001484. PMID 27661661
- [Background] Barbado J, Tabera S, Sanchez A, Garcia-Sancho J. Therapeutic potential of allogeneic mesenchymal stromal cells transplantation for lupus nephritis. Lupus. 2018 Nov;27(13):2161-2165. doi: 10.1177/0961203318804922. Epub 2018 Oct 5. PMID 30290717
- [Background] Leng Z, Zhu R, Hou W, Feng Y, Yang Y, Han Q, Shan G, Meng F, Du D, Wang S, Fan J, Wang W, Deng L, Shi H, Li H, Hu Z, Zhang F, Gao J, Liu H, Li X, Zhao Y, Yin K, He X, Gao Z, Wang Y, Yang B, Jin R, Stambler I, Lim LW, Su H, Moskalev A, Cano A, Chakrabarti S, Min KJ, Ellison-Hughes G, Caruso C, Jin K, Zhao RC. Transplantation of ACE2- Mesenchymal Stem Cells Improves the Outcome of Patients with COVID-19 Pneumonia. Aging Dis. 2020 Mar 9;11(2):216-228. doi: 10.14336/AD.2020.0228. eCollection 2020 Apr. PMID 32257537